CLINICAL TRIAL: NCT02833038
Title: Effect of Intravenous Magnesium During Robot Assisted Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Ji Eun Kim, Assistant professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AJIRB-MED-CT4-16-074
Record Dates: First submitted 2016-07-12; First posted 2016-07-14 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnesium Sulfate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Magnesium group (Experimental): Intravenous administration of Magnesium Sulfate
  Interventions: Drug: Magnesium Sulfate
- Control group (Placebo Comparator): Intravenous administration of normal saline
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Magnesium Sulfate — adminstration of intravenous magnesium as bolus of 50 mg/kg, followed by continuous infusion at rate of 10 mg/kg/h
  Arms: Magnesium group
Drug: Normal saline — the same bolus and infusion volumes of normal saline
  Arms: Control group

SUMMARY:
The primary purpose of this study is to investigate the effect of intravenous magnesium on blood pressure after Trendelenburg position during robot assisted prostatectomy.

The secondary purpose of this study is to investigate the effect of intravenous magnesium on pain after robot assisted prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Robot assisted prostatectomy

Exclusion Criteria:

* Allergy to magnesium
* Chronic pain
* Chronic opioid use
* Chronic NSAID use
* Renal dysfunction
* Liver dysfunction
* Cardiac arrythmia
* Seizure

Ages: 60 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Mean blood pressure | Up to 2 hours after Trendelenburg position

SECONDARY OUTCOMES:
Postoperative pain | Up to 24 hours after surgery end
  pain assessment using visual analog scale

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Ajou University School of Medicine, Suwon, Seoum, South Korea

REFERENCES:
- [Derived] Kim HY, Lee SY, Lee HS, Jun BK, Choi JB, Kim JE. Beneficial Effects of Intravenous Magnesium Administration During Robotic Radical Prostatectomy: A Randomized Controlled Trial. Adv Ther. 2021 Mar;38(3):1701-1712. doi: 10.1007/s12325-021-01643-8. Epub 2021 Feb 21. PMID 33611742